CLINICAL TRIAL: NCT00492583
Title: Study to Investigate the Potential of Probiotics in Yogurt
Acronym: SIPPY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Daniel Merenstein, Georgetown University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2007-273
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: probiotic; health; bifidobacterium lactis; BB-12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects were provided 4 fluid ounces (112 grams) administered orally per day of placebo drink.
  Interventions: Drug: Placebo
- Bifidobacterium lactis (BB-12) (Experimental): Subjects were provided 4 fluid ounces (112 grams) administered orally per day of active drink.
  Interventions: Drug: Bifidobacterium lactis (BB-12)

INTERVENTIONS:
Drug: Bifidobacterium lactis (BB-12) — The active drink is currently available commercially on campus at The Berkey Creamery at Penn State in State College, Pennsylvania. The active drink combined a commercial blend (YFL-702, Chr.) of the following active cultures, Streptococcus thermophilus and Lactobacillus delbrueckii subsp. bulgaricus. The active drink was also supplemented with the probiotic BB-12, acquired from Chr. Hansen (Milwaukee, Wisconsin).
  Arms: Bifidobacterium lactis (BB-12)
Drug: Placebo — The placebo drink combined a commercial blend (YFL-702, Chr.) of the following active cultures, Streptococcus thermophilus and Lactobacillus delbrueckii subsp. bulgaricus.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the consumption of a yogurt drink containing a high dose of probiotics decreases absences, due to illnesses, in daycare centers for children between the ages of 1 and 3.

DETAILED DESCRIPTION:
It is reported that more than half of all young children attend daycare centers in the United States. Absences due to illnesses are costly both on an individual and societal level; these absences are generally due to diarrhea or upper respiratory infections.

In the U.S., children under five years of age experience 20-35 million episodes of diarrhea per year. These episodes lead to 2-3.5 million physician visits (which account for 10% of all visits by children), more than 200,000 hospitalizations (13% of hospital admissions in children under five years), and 325-425 deaths annually. In 1991, the outpatient costs of treating diarrhea in children under age three was calculated at 0.6-1 billion dollars per year.

Respiratory illness is among the leading causes of death in children under five years of age. Approximately 200,000 deaths in the U.S. and 3.9 million deaths worldwide are attributed to respiratory illnesses. Respiratory illness is also the most frequent reason for physician consultation, with more than 40% of all pediatric outpatient visits related to respiratory illness. According to a recent study, 39% of children attending daycare experienced acute otitis media (ear infection) and 26% reported allergies. Most notably, 10% of children attending daycare were admitted to the hospital due to respiratory illnesses.

We have chosen BB-12 as the probiotic for this study as it is one of the best characterized probiotics with a long safety record in children, a well-proven ability to colonize the human intestinal tract, and demonstrated efficacy for different pediatric conditions. Furthermore, BB-12 is a commercially available probiotic strain that has been used in a number of feeding and clinical trials.

In fact, there is a new infant formula on the market, using the identical strain we are, in the first commercially available probiotic infant formula available in the United States. Not only has BB-12 been found to survive transit through the stomach, small intestine and colon, but also long-term consumption of BB-12 formula at levels as high as 1 billion CFU/g (240 g serving) have been found to be safe.

Our overall goal is to demonstrate that a probiotic-containing yogurt beverage can be used successfully as a vehicle for delivering health-enhancing probiotics; more specifically to determine if a yogurt drink containing Bifidobacterium lactis BB-12 at a minimum 1010 colony forming units (CFU)/per serving can prevent daycare absences.

The rationale for focusing on food as a vehicle for the transmission of probiotics is that it has the potential to benefit children more than using probiotics in a more medicinal manner, such as pills or capsules. By providing an intervention in the form of a yogurt drink, parents are given a more convenient and simple alternative to traditional probiotic supplements. As yogurt is known to be a nutrient dense food, a yogurt drink is likely to be more appealing to both children and their parents for long-term consumption than pharmaceutical-like preparations. Although compliance with most medicinal regimens is around 50%, by offering a more attractive formulation of high dose probiotics and collaborating with participants we believe compliance will exceed normal levels. Ultimately, by capitalizing on the widely accepted healthy image of yogurt and offering a simple, convenient source of probiotics, we believe this product has the potential to positively impact the health of children around the world.

ELIGIBILITY:
Inclusion Criteria:

* aged 1-3
* attending daycare or preschool centers at least 3 days a week
* male or female
* parents must speak English or Spanish
* subjects or parents/legal guardians who agree to have their child refrain from consuming any other yogurts or foods containing probiotics for the duration of the study

Exclusion Criteria:

* subjects with developmental delays
* subjects with chronic conditions such as diabetes or asthma that require daily medication
* subjects with birth weight <2500 grams
* subjects with strawberry allergies
* subjects with active diarrhea
* subjects with congenital anomalies
* subjects with failure to thrive
* subjects with parental belief of lactose intolerance

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Merenstein, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Department of Family Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Merenstein DJ, Smith KH, Scriven M, Roberts RF, Sanders ME, Petterson S. The study to investigate the potential benefits of probiotics in yogurt, a patient-oriented, double-blind, cluster-randomised, placebo-controlled, clinical trial. Eur J Clin Nutr. 2010 Jul;64(7):685-91. doi: 10.1038/ejcn.2010.30. Epub 2010 Mar 10. PMID 20216564

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Bifidobacterium Lactis (BB-12)
Started | 95 | 87
Completed | 95 | 87
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bifidobacterium Lactis (BB-12) | Total
Number analyzed (Participants) | 95 | 87 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 95 | 87 | 182
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 36 | 43 | 79
  Male | 50 | 34 | 84
  Missing | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 95 | 87 | 182

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Children Are Out of School Sick
Description: Outcome measure, "number of days children are out of school sick" was measured for the entire population
Time Frame: 90 days
Measure: Number; unit: days per 100 person days
Arm/Group | Placebo | Bifidobacterium Lactis (BB-12)
Number analyzed (Participants) | 95 | 87
days per 100 person days | 2.51 | 2.82

ADVERSE EVENTS:
Arm/Group | Placebo | Bifidobacterium Lactis (BB-12)
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/87
Other Adverse Events (participants affected / at risk) | 3/95 | 3/87
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=95) | Bifidobacterium Lactis (BB-12) (N=87)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Dermatitis (Diaper) (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Vomiting & Cough (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hordeolum (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No